CLINICAL TRIAL: NCT04732429
Title: A Phase 2 Open-label, Dose Escalation Study of HST5040 in Subjects With Propionic or Methylmalonic Acidemia Followed by a Randomized, Double-blind, Placebo-controlled, 2-period Crossover Study and an Open-label, Long-term Extension Study
Brief Title: Study of HST5040 in Subjects With Propionic or Methylmalonic Acidemia
Acronym: HERO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to terminate the study was based on business considerations by the Sponsor.
Sponsor: HemoShear Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HST20-CL01
Record Dates: First submitted 2021-01-21; First posted 2021-02-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Methylmalonic Acidemia; Propionic Acidemia
Keywords: Methylmalonic Acidemia; Propionic Acidemia; Organic Acidemia; Inborn errors of metabolism; PCCA; PCCB; Propionyl-coenzyme A carboxylase; MMUT; Methylmalonyl-CoA mutase; Metabolic disease; Genetic disease; HemoShear
MeSH Terms: conditions — Methylmalonic acidemia; Propionic Acidemia; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Drug (Experimental): Part B is the 6-month, randomized, double-blind (Subject/Investigator/Sponsor), placebo-controlled, 2-period crossover study consisting of 2 intervention periods of 12 weeks each to evaluate the safety and efficacy of the optimal dose of HST5040 in PA and MMA subjects ≥ 2 years old (N = minimum 12) in addition to SoC determined in Part A (within-subject dose escalation).
  Interventions: Drug: HST5040
- Placebo (Experimental): Placebo in addition to standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HST5040 — Liquid solution
  Arms: Active Drug
Drug: Placebo — Liquid solution
  Arms: Placebo

SUMMARY:
This is an interventional study to assess the safety, PK, and efficacy of HST5040 in 12 subjects - 6 with Methylmalonic Acidemia (MMA) and 6 with Propionic Acidemia (PA). The study consists of 3 parts:

* Part A: Open-label, within-subject, dose escalation study in PA and MMA subjects ≥ 2 years old to identify a safe and pharmacologically active (optimal) dose of HST5040 for use in Part B. Subjects will continue in a Part A open-label extension until all subjects complete Part A and the optimal dose of HST5040 is identified for use in Part B.
* Part B: 6-month, randomized, double-blind, placebo-controlled, 2-period crossover in the same subjects from Part A to evaluate safety and efficacy of the optimal dose of HST5040 in addition to standard of care (SoC).
* Part C: open-label long-term extension study in PA and MMA subjects ≥ 2 years old (N = approximately 12, 6 each) to evaluate the long-term safety and efficacy of the optimal dose of HST5040.

This study will determine whether HST5040 can improve levels of disease-associated toxins that accumulate in patients with PA and MMA.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of symptomatic PA or MMA (Mutase)
* Ages ≥ 2 years old.
* History of Inadequate metabolic control while receiving standard of care (SoC).
* Plasma MCA concentration > 3x upper limit of normal of the reference range at screening.
* Stable supplementation dose of carnitine for at least 1 week prior to the entry in the study.

Exclusion Criteria:

* Moderate-to-severely impaired cardiac function with LVEF < 45% by ECHO.
* Clinically significant arrhythmia by Holter monitor.
* QTcF > 450 msec
* Moderate to severe chronic kidney disease with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2.
* Exposure to any investigational therapy, apart for a COVID-19 vaccine, within the past 6 months prior to study entry.
* Exposure to gene therapy for PA or MMA at any time prior to study entry.
* History of organ transplantation (Part A and B only)
* History of severe allergic or anaphylactic reactions to any of the components of HST5040.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change in plasma 2-methylcitric acid (MCA) levels | 6 months
  nmol/mL

SECONDARY OUTCOMES:
Change in plasma propionyl-carnitine (3) | 6 months
  µmol/L
Change in C3 to acetyl-carnitine ratio (C3:C2) | 6 months
  µmol/L
Change in 3-OH propionate | 6 months
  g/mol
Change in Methylmalonic acid (in MMA subjects) | 6 months
  nmol/L
Change in NH3 | 6 months
  nmol/L
Anion Gap | 6 months
  mEq/L
Pharmacokinetics parameters - Cmax | 6 months
  Maximum concentration (Cmax) after administration of HST5040
Pharmacokinetics parameters - Tmax | 6 months
  Time of maximum concentration (Tmax)
Pharmacokinetics parameters - AUC | 6 months
  Area under the concentration time curve (AUC)
Oral Intake | 6 months
  Food diary - change from baseline to end of each dose level interval in oral intake
Acute Metabolic Decompensations | 6 months
  Change in the total number of metabolic decompensation events requiring an emergency room (ER) visit of hospitalization
MetabQoL 1.0 - Health Related Quality of Life (HRQOL) | 6 months
  Score 0-100 Scale. Higher Score indicates better HRQOL
PedsQL 1.0 Family Impact Score - Health Related Quality of Life (HRQOL) | 6 months
  Score 0-100 Scale. Higher Score indicates better HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Horn, MD PhD, Study Chair — HemoShear Therapeutics, Inc.
Locations (16):
- United States (14):
  - Rady Children's Hospital, San Diego, California
  - Yale, New Haven, Connecticut
  - Children's National Health System, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - John P. and Kathrine G. McGovern Medical School, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- King Faisal Specialist Hospital and Research Centre, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No